CLINICAL TRIAL: NCT00649844
Title: Double Blind, Double-Dummy Multicenter, Parallel Group Comparison Of The Efficacy And The Tolerability Of Ziprasidone Vs. Clozapine In Schizophrenic Patients Who Are Refractory And/Or Intolerant To Antipsychotic Therapy
Brief Title: A Study Comparing the Efficacy and Tolerability of Ziprasidone vs. Clozapine for the Treatment of Schizophrenia in Patients Who Continue to Have Symptoms on or Cannot Tolerate Other Antipsychotic Drugs
Acronym: MOZART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1281039
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Clozapine; ziprasidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Clozapine
- B (Experimental)
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Clozapine — Clozapine 25 or 100 mg tablets. Patients were initially titrated over the first 10 days to 300 mg/day and remained at this dose for 1 week. Thereafter, the dose could be varied between 250 and 600 mg/day based on response and tolerability for a total treatment duration of 18 weeks
  Arms: A
Drug: Ziprasidone — Ziprasidone 40, 60, or 80 mg capsules. Patients were initially titrated over the first 3 days to 80 mg/day, which could subsequently be increased to between 80 and 160 mg/day based on response and tolerability for a total treatment duration of 18 weeks
  Other Names: Geodon, Zeldox
  Arms: B

SUMMARY:
The purpose of this study is to compare the efficacy and safety of ziprasidone and clozapine in schizophrenic patients who are resistant and/or intolerant to antipsychotic treatment

ELIGIBILITY:
Inclusion Criteria:

* CGI - S ≥4
* PANSS ≥ 80
* Inpatients or outpatients

Exclusion Criteria:

* Patients with a history of myeloproliferative diseases, history of granulocytopenia, agranulocytosis due to a drug
* Diagnosis of substance dependence within previous 3 months using DSM-IV criteria
* History of seizure
* Organic mental disease, including mental retardation or epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2003-01; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline to endpoint in Positive and Negative Syndrome Scale (PANSS) total scores | Until Final Visit (within 18 weeks)

SECONDARY OUTCOMES:
Proportion of responders, based on change from baseline to endpoint in PANSS total score | Until Final Visit (within 18 weeks)
Change from baseline to endpoint in Clinical Global Impressions-Severity (CGI-S) scores | Baseline and weekly from Weeks 1-18
Time to discontinuation | Up to 18 weeks
Change from baseline to endpoint in cognitive function assessments, including Rey serial verbal learning test, Stroop Color Word test, and Trail Making Test | Baseline and Weeks 12 and 18
Change from baseline to endpoint in Global Assessment of Functioning (GAF) scores | Baseline and Week 8, 12, and 18
Change from baseline in Modified Resource Utilization Questionnaire (RUQ) scores | Baseline and Weeks 4, 8, 12, and 18
Change from baseline to endpoint in Drug Attitude Inventory (DAI) scores | Screening and Weeks 1, 8, 12, and 18
Change from baseline to endpoint in PANSS subscale scores | Baseline and weekly from Weeks 1-18
Adverse events | Weekly from Weeks 1-18
Change from baseline to endpoint in Calgary Depression Scale (CDSS) scores | Baseline and Weeks 8, 12, and 18
Change from baseline in Caregiver Activity Survey (CAS) | Screening and Weeks 1, 8, 12, and 18
Change from baseline in laboratory tests | Screening and weekly from Weeks 1-18
Change from baseline in electrocardiogram | Screening and Weeks 1, 8, 12, and 18
Change from baseline in movement disorder rating scales, including Barnes Akathisia Rating Scale, Abnormal Involuntary Movement Scale, and Simpson-Angus Scale | Baseline and Weeks 1, 8, 12, and 18
Change from baseline to endpoint in Clinical Global Impressions-Improvement (CGI-I) scores | Baseline and weekly from Weeks 1-18
Change from baseline to endpoint in Patient Preference Scale (PPS) scores | Screening and Weeks 1, 8, 12, and 18

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- Italy (19):
  - Pfizer Investigational Site, Città di Castello, Perugia
  - Pfizer Investigational Site, Bassano del Grappa, Vicenza
  - Pfizer Investigational Site, Bari
  - Pfizer Investigational Site, Brescia
  - Pfizer Investigational Site, Cagliari
  - Pfizer Investigational Site, Catania
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Guardiagrele (CH)
  - Pfizer Investigational Site, Messina
  - Pfizer Investigational Site, Montichiari (brescia)
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Parma
  - Pfizer Investigational Site, Reggio Calabria
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Sassari
  - Pfizer Investigational Site, Siena
  - Pfizer Investigational Site, Torino
  - Pfizer Investigational Site, Trieste
  - Pfizer Investigational Site, Verona
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281039&StudyName=A%20study%20comparing%20the%20efficacy%20and%20tolerability%20of%20ziprasidone%20vs.%20clozapine%20for%20the%20treatment%20of%20schizophrenia%20in%20patients%20who%20continue